CLINICAL TRIAL: NCT02776072
Title: A Multicenter, Global, Retrospective, Observational Study to Characterize Real-world Clinical Outcomes in Patients With Relapsing-remitting Multiple Sclerosis Treated With Disease-modifying Therapies (Tecfidera®, Copaxone®, Aubagio®, or Gilenya®)
Brief Title: Observational Study to Characterize Real-world Clinical Outcomes With Relapsing-remitting Multiple Sclerosis (RRMS)
Acronym: EFFECT
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: 109MS421
Record Dates: First submitted 2016-05-16; First posted 2016-05-18 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Multiple Sclerosis
Keywords: Tecfidera, DMF, dimethyl fumarate, Fingolimod, Glatiramer acetate, Teriflunomide, Gilenya, Copaxone, Aubagio
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- dimethyl fumarate (DMF): Participants who initiated DMF during the specified time period
- glatiramer acetate (GA): Participants who initiated GA during the specified time period
- teriflunomide: Participants who initiated teriflunomide during the specified time period
- fingolimod: Participants who initiated fingolimod during the specified time period

SUMMARY:
The primary objective of the study is to evaluate the real-world clinical effectiveness, as measured by the proportion of participants relapsed at 12 months, in participants treated with dimethyl fumarate (DMF).

Secondary objectives of the study are: To evaluate the real-world clinical effectiveness, as measured by the proportion of participants relapsed at 12 months, in participants treated with DMF, glatiramer acetate (GA), teriflunomide, or fingolimod both in the overall participant cohort and in a subset of participants who were naïve to disease-modifying therapy (DMT) and were diagnosed with multiple sclerosis (MS) within 3 years of starting the index therapy; To compare relapse activity, defined as annualized relapse rate (ARR), among participants treated with DMF, GA, teriflunomide, or fingolimod; To compare MS-related hospitalizations among participants treated with DMF, GA, teriflunomide, or fingolimod; To compare intravenous corticosteroid use among participants treated with DMF, GA, teriflunomide, or fingolimod.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of RRMS per McDonald criteria
* Initiated treatment with DMF, GA, teriflunomide, or fingolimod (defined as index therapy) no earlier than January 2011 and no later than 12 months prior to the date of medical record abstraction (i.e., patient has at least 12 months of data available in the medical record following initiation of index treatment). Note: Patients who have initiated the index therapy but subsequently discontinued or switched to other therapies are allowed in this study as long as there is at least 12 months of follow-up following the initiation of the index therapy.
* Have sufficient available medical records for data abstraction to meet the objectives of the study, i.e., the patient was either under the medical care of the investigating site during the entire period of the index treatment or the patient's complete MS disease and treatment history is otherwise available at the investigating site

Key Exclusion Criteria:

* Diagnosis of a progressive form of MS (progressive relapsing, primary progressive, secondary progressive) at any time before or during the period for which data will be collected
* Have received disease-modifying therapies other than one platform therapy (IFN or GA) prior to initiation of index therapy. In patients for whom GA is index therapy, only one prior IFN therapy is allowed.
* Have received any formulations of DMF, Fumaderm®, or compounded fumarates (e.g., Psorinovo) at any time prior to initiation of treatment with Tecfidera®
* Concurrent enrollment in any interventional clinical trial of an investigational product during time evaluated for medical record abstraction

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with a diagnosis of RRMS treated with dimethyl fumarate, fingolimod, teriflunomide, or glatiramer acetate in routine clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 2978 (Actual)
Dates: Start 2016-05; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Proportion of participants relapsed at 12 months in participants treated with DMF | One day
  Single time point per participant retrospective medical record abstraction with no required study visits or procedures

SECONDARY OUTCOMES:
Proportion of participants relapsed at 12 months treated with index therapy in the overall population as well as the subgroup of MS participants who were naïve to DMTs and were diagnosed with MS within 3 years of starting the index therapy | One day
  Single time point per participant retrospective medical record abstraction with no required study visits or procedures
ARR at 12 months in participants treated with index therapy in the overall population as well as in the matched cohorts | One day
  Single time point per participant retrospective medical record abstraction with no required study visits or procedures
Proportion of relapsed participants with one or more MS-related hospitalizations during the 12 months following treatment initiation in participants treated with index therapy in the overall population and the matched cohorts | One day
  Single time point per participant retrospective medical record abstraction with no required study visits or procedures
Proportion of relapsed participants requiring treatment with intravenous corticosteroids during the 12 months following treatment initiation in participants treated with index therapy in the overall participant population and the matched cohorts | One day
  Single time point per participant retrospective medical record abstraction with no required study visits or procedures

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (114):
- United States (36):
  - Research Site, Homewood, Alabama
  - Research Site, Gilbert, Arizona
  - Research Site, Hanford, California
  - Research Site, Modesto, California
  - Research Site, Santa Ana, California
  - Research Site, Aurora, Colorado
  - Research Site, Danbury, Connecticut
  - Research Site, Hartford, Connecticut
  - Research Site, Jacksonville, Florida
  - Research Site, Port Orange, Florida
  - Research Site, Savannah, Georgia
  - Research Site, Avon, Indiana
  - Research Site, Franklin, Indiana
  - Research Site, Muncie, Indiana
  - Research Site, Overland Park, Kansas
  - Research Site, Boston, Massachusetts
  - Research Site, Wellesley, Massachusetts
  - Research Site, Golden Valley, Minnesota
  - Research Site, Amherst, New York
  - Research Site, New Hyde Park, New York
  - Research Site, New York, New York
  - Research Site, Patchogue, New York
  - Research Site, Raleigh, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Medford, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Dallas, Texas
  - Research Site, Houston, Texas
  - Research Site, Mansfield, Texas
  - Research Site, Round Rock, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Norfolk, Virginia
  - Research Site, Tacoma, Washington
- Argentina (5):
  - Research Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Research Site, Ciudad Autonoma Buenos Aires, Ciudad Autonoma Buenos Aires
  - Research Site, Córdoba, Córdoba Province
  - Research Site, Salta, Salta Province
  - Research Site, Rosario, Santa Fe Province
- Australia (4):
  - Research Site, New Lambton Heights, New South Wales
  - Research Site, Box Hill, Victoria
  - Research Site, Heidelberg, Victoria
  - Research Site, Melbourne, Victoria
- Canada (8):
  - Research Site, Burnaby, British Columbia
  - Research Site, Saint John, New Brunswick
  - Research Site, Halifax, Nova Scotia
  - Research Site, Cambridge, Ontario
  - Research Site, Guelph, Ontario
  - Research Site, Chicoutimi, Quebec
  - Research Site, Gatineau, Quebec
  - Research Site, Greenfield Park, Quebec
- Croatia (2):
  - Research Site, Osijek
  - Research Site, Varaždin
- Czechia (8):
  - Research Site, Brno
  - Research Site, Hradec Králové
  - Research Site, Jihlava
  - Research Site, Olomouc
  - Research Site, Ostrava-Poruba
  - Research Site, Pardubice
  - Research Site, Prague
  - Research Site, Teplice
- France (4):
  - Research Site, Libourne, Gironde
  - Research Site, Toulouse, Haute Garonne
  - Research Site, Le Mans, Sarthe
  - Research Site, Le Chesnay, Yvelines
- Germany (21):
  - Research Site, Freiburg im Breisgau, Baden-Wurttemberg
  - Research Site, Pforzheim, Baden-Wurttemberg
  - Research Site, Stuttgart, Baden-Wurttemberg
  - Research Site, Bamberg, Bavaria
  - Research Site, Potsdam, Brandenburg
  - Research Site, Hamburg, Hamburg
  - Research Site, Kassel, Hesse
  - Research Site, Oldenburg, Lower Saxony
  - Research Site, Osnabrück, Lower Saxony
  - Research Site, Stade, Lower Saxony
  - Research Site, Bochum, North Rhine-Westphalia
  - Research Site, Düsseldorf, North Rhine-Westphalia
  - Research Site, Gelsenkirchen, North Rhine-Westphalia
  - Research Site, Hagen, North Rhine-Westphalia
  - Research Site, Siegen, North Rhine-Westphalia
  - Research Site, Sprockhövel, North Rhine-Westphalia
  - Research Site, Kandel, Rhineland-Palatinate
  - Research Site, Saint Ingbert, Saarland
  - Research Site, Leipzig, Saxony
  - Research Site, Kiel, Schleswig-Holstein
  - Research Site, Berlin, State of Berlin
- Hungary (6):
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Eger
  - Research Site, Esztergom
  - Research Site, Kecskemét
  - Research Site, Nyíregyháza
- Italy (3):
  - Research Site, Cagliari, Cagliari
  - Research Site, Catania, Catania
  - Research Site, Napoli, Napoli
- Spain (8):
  - Research Site, Alicante, Alicante
  - Research Site, Badalona, Barcelona
  - Research Site, Córdoba, Cordoba
  - Research Site, Santiago de Compostela, La Coruña
  - Research Site, Madrid, Madrid
  - Research Site, Málaga, Malaga
  - Research Site, Vigo, Pontevedra
  - Research Site, Seville, Sevilla
- Switzerland (2):
  - Research Site, Lausanne
  - Research Site, Lugano
- United Kingdom (7):
  - Research Site, Truro, Cornwall
  - Research Site, Exeter, Devon
  - Research Site, Chelmsford, Essex
  - Research Site, Romford, Essex
  - Research Site, London, Greater London
  - Research Site, Glasgow, Strathclyde
  - Research Site, Chertsey, Surrey

REFERENCES:
- [Derived] Min J, Cohan S, Alvarez E, Sloane J, Phillips JT, van der Walt A, Koulinska I, Fang F, Miller C, Chan A. Real-World Characterization of Dimethyl Fumarate-Related Gastrointestinal Events in Multiple Sclerosis: Management Strategies to Improve Persistence on Treatment and Patient Outcomes. Neurol Ther. 2019 Jun;8(1):109-119. doi: 10.1007/s40120-019-0127-2. Epub 2019 Jan 31. PMID 30706431